CLINICAL TRIAL: NCT01643486
Title: Development of a 'Phosphate Counting Program' on an iTouch to Simplify Self-management of Dietary Phosphate by Patients With End Stage Renal Disease(ESRD) Treated With Peritoneal Dialysis
Brief Title: Development of a 'Phosphate Counting Program'
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Baxter Healthcare Corporation (Industry); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iTouch Phase 3
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: End Stage Renal Disease
Keywords: peritoneal dialysis; phosphate; iTouch
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- iTouch phosphate counting program (Experimental): All patients will have an iTouch that will help them to calculate the required number of phosphate binders to be taken with each meal
  Interventions: Other: iTouch phosphate counting program
- Usual Care (Active Comparator): Participants in the active comparator group will document their meals in the iTouch but continue to take their phosphate binders as prescribed by their MD/dietician
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: iTouch phosphate counting program — After developing and pilot testing the iTouch phosphate counting program, the participants in the intervention arm will enter their meal into the program; the required number of phosphate binders will be calculated for the patient
  Arms: iTouch phosphate counting program
Other: Usual Care — The patients randomized to the usual care arm will continue to receive the usual dietary counselling and will input meal data into the iTouch program but no recommendations for the number of phosphate binders to be taken with the meal will be provided
  Arms: Usual Care

SUMMARY:
Hypothesis: The use of a program that assists with selection of the appropriate number of phosphate binders for a meal based on patient specific factors will result in improved serum phosphate control, a reduction in overall number of phosphate binders used and enhanced patient satisfaction.

Primary Aim: To determine if teaching patients to use a 'phosphate counting' program installed on an iTouch that selects the appropriate amount of phosphate binder to be taken with each meal is associated with better phosphate control than usual care.

Research Plan: There will be 3 phases to the study. Phase 1: Recruitment of 60 peritoneal dialysis (PD) patients. The information generated from this phase will be used to develop the iTouch program for phosphate counting and matching binder number. Phase 2: iTouch program once developed will be pilot tested on a convenience sample of 10 PD patients and modified if required. Phase 3: Randomized controlled trial of 92 PD patients to determine if using the iTouch phosphate counting program reduces serum phosphate compared to controls. Success would be based on seeing a statistically significant difference in serum phosphate as expected from our sample size calculation

DETAILED DESCRIPTION:
Project approach and work plan:

Phase 1: In the week prior to the collection of standard pre-clinic blood work (to include calcium, phosphate, PTH), PD patients will keep a 3-day diary that will include all foods and beverages consumed in addition to the portion sizes. At the time of standard pre-clinic bloodwork collection, patients will perform an adequest. Medication lists will be reviewed for: 1) Proton pump inhibitors/ H2 receptor antagonists 2) 25-hydroxyvitamin D3 and 1,25 dihydroxyvitamin D3 and 3) phosphate binders. Doses taken the week prior to standard pre-clinic blood work when the diet diaries are compiled will be recorded. This information will be used for 2 separate purposes: 1) A list of the foods that are actually being eaten by the PD patients will be generated 2) The 3-day average phosphate content will be estimated from each PD patient's food diaries. A regression equation that predicts serum phosphate concentration taking into account phosphate intake, the amount of phosphate binders taken, the dose of vitamin D, use of proton pump inhibitors/H2 antagonists, dialysis adequacy, and serum PTH concentration will be generated.

Phase 2: An iTouch program will be developed using Phase 1 information to assist patients in meal phosphate counting and appropriate binder selection. Processes used to develop similar programs such as the pilot study in patients with diabetes mellitus will be used. A convenience sample of 10 PD patients will use the iTouch program for one month and document their impressions about ease of use, convenience and applicability to their diet choices. Changes to the program will be incorporated based on the patient's comments and laboratory values. If substantial changes are required, another convenience sample of 10 PD patients will be invited to use the program and provide feedback.

Phase 3: 80 consenting PD patients from the Ottawa Hospital and St. Michael's Hospital (if required) will be randomized to usual care for managing phosphate versus use of the iTouch program for meal phosphate counting and matching binder use. This phase of the trial will last 3 months. As simply recording meal phosphate intake in the iTouch program may have an impact on patient behavior, the control group will be asked to enter this data into the program but no binder therapy information will be provided to the patients. During the course of the study, the dose of vitamin D and PD prescription will be held constant in both groups.

Expected Outcome:

Phase 1: All 60 PD patients will be recruited over a 6-month period. Data entry and statistical analysis are expected to take another 2-4 months. Phase 2: Actual development of the iTouch program using the data generated in phase 1 is expected to take about 6 months. It is anticipated that all 10 patients will be recruited over a 2-month period with a further one-month of follow-up. Interviews with the patients and collation of the data are expected to take another month. It is unclear how much time will be required to make adjustments to the iTouch program but we anticipate <3months.

Phase 3: We anticipate that we can recruit the 80 patients from the greater than 250 patients at the Ottawa Hospital and St Michaels Home Dialysis programs and complete the 3 months of follow-up in approximately 12-18months. Data analysis and manuscript preparation should take another 4-5 months.

Feasibility Given the large number of PD patients in the two programs, the novelty of Phase 2 and 3 and the incentives in Phase 3, we do not anticipate difficulties with recruitment. The laboratory tests are all standard and visits will occur during a patient's regularly scheduled PD visit.

ELIGIBILITY:
Inclusion Criteria:

1. End stage renal disease treated with peritoneal dialysis
2. On calcium carbonate phosphate binder therapy
3. English or French speaking/writing

Exclusion Criteria:

1. Cognitive dysfunction that might interfere with ability to participate
2. Unable or unwilling to give informed consent
3. Hypercalcemia
4. Visually impaired
5. Hearing impaired
6. Expected renal transplant during the time of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Serum Phosphate | 3 months
  The primary end point of the study will be a comparison of the serum phosphate between the two study groups at the end of the 3 months. An unpaired t-test will be used with a value of <0.05 considered to be statistically significant in an intent to treat analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farfan-Ruiz AC, Czikk D, Leidecker J, Ramsay T, McCormick B, Wilson K, Zimmerman D. Multidisciplinary Team versus a "Phosphate-Counting" App for Serum Phosphate Control: A Randomized Controlled Trial. Kidney360. 2020 Dec 15;2(2):290-297. doi: 10.34067/KID.0007132020. eCollection 2021 Feb 25. PMID 35373021